CLINICAL TRIAL: NCT01771614
Title: The Effects of Hyperglycaemia on the Response to Acute Exercise
Brief Title: Glucotoxicity and Acute Exercise
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated to a different country.
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GlucotoxEx
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Glucotoxicity; Exercise; Beta-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normoglycemia + exercise (Experimental): At T = 0 h participants will undergo an intravenous glucose tolerance test (IVGTT, 0.33 g/kg glucose) immediately followed by a 4-hour rest period. At T = 5 h, participants will undertake 45 minutes of moderate-intensity (70% VO2max) bicycle ergometry. Immediately following (T = 6 h) and 1- (T = 7 h), 3- (T = 9 h), and 18- hours (T = 24 h) after exercise, participants will undergo additional IVGTTs.
  Interventions: Behavioral: Exercise
- Steady-State Hyperglycemia + exercise (Experimental): At T = 0 h participants will undergo an intravenous glucose tolerance test (IVGTT, 0.33 g/kg glucose) immediately followed by a 4-hour rest period. During this time, steady-state hyperglycemia (~10 mM) will be induced experimentally via a variable-rate intravenous infusion of 20% dextrose. At T = 5 h, participants will undertake 45 minutes of moderate-intensity (70% VO2max) bicycle ergometry. Immediately following (T = 6 h) and 1- (T = 7 h), 3- (T = 9 h), and 18- hours (T = 24 h) after exercise, participants will undergo additional IVGTTs.
  Interventions: Behavioral: Exercise; Procedure: Hyperglycemia
- Fluctuating Hyperglycemia + exercise (Experimental): At T = 0 h participants will undergo an intravenous glucose tolerance test (IVGTT, 0.33 g/kg glucose) immediately followed by a 4-hour rest period. During this time, fluctuating hyperglycemia (~8-15 mM) will be induced by intravenously injecting 0.15 g/kg boluses of 20% dextrose every 30 minutes. At T = 5 h, participants will undertake 45 minutes of moderate-intensity (70% VO2max) bicycle ergometry. Immediately following (T = 6 h) and 1- (T = 7 h), 3- (T = 9 h), and 18- hours (T = 24 h) after exercise, participants will undergo additional IVGTTs.
  Interventions: Behavioral: Exercise; Procedure: Hyperglycemia

INTERVENTIONS:
Behavioral: Exercise
Procedure: Hyperglycemia
  Arms: Fluctuating Hyperglycemia + exercise; Steady-State Hyperglycemia + exercise

SUMMARY:
Experimental hyperglycemia (5 hours) will be induced via a constant- or fluctuating-rate glucose infusion to establish different patterns of glycemia in healthy individuals. The effects of these acute models of hyperglycemia on the adaptations to a single aerobic exercise bout will be tested. Changes in pancreatic endocrine function, insulin sensitivity, endothelial function, and oxidative stress will be measured.

ELIGIBILITY:
Inclusion criteria for participation:

* Male
* Age 18-50 years
* Body Mass Index 19-30 kg/m2
* Generally healthy

Exclusion criteria for participation:

* Regular use of anti-inflammatory medication
* Smokers
* More than 2 kg weight change in prior 6 months
* Previous weight loss surgery
* Cancer, or evidence of chronic haematological, pulmonary, cardiac, hepatic, renal, or gastrointestinal disease
* Evidence of diabetes
* Engaged in moderate or vigorous activity on more than 5 days per week

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Estimated); Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Pancreatic endocrine function | 0, 6, 7, 9, and 24 hours
  The plasma insulin, C-peptide, and glucagon responses to a 0.33 g/kg intravenous glucose tolerance test (IVGTT) will be measured. In each trial, the IVGTT will be performed at T = 0, 6, 7, 9, and 24 hours.

SECONDARY OUTCOMES:
Glucose tolerance | 0, 6, 7, 9, and 24 hours
  Glucose tolerance will be measured during an IVGTT in each trial at T = 0, 6, 7, 9, and 24 hours.
Endothelial function | 0, 6, 7, 9, and 24 hours
  Blood flow and flow-mediated dilation by Doppler ultrasound will be measured in each trial at T = 0, 6, 7, 9, and 24 hours.
Oxidative stress | 24 hours
  Urine will be collected over the whole 24-hour period of each trial and 8-iso Prostaglandin F3α will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom